CLINICAL TRIAL: NCT00301912
Title: Phase II Study Evaluating Busulfan and Fludarabine as Preparative Therapy in Adults With Hematopoietic Disorders Undergoing Matched Unrelated Donor Stem Cell Transplantation
Brief Title: Busulfan and Fludarabine Before Donor Stem Cell Transplant in Treating Patients With Hematologic Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn because study never opened to accrual
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Thomas G. Martin, III, UCSF Helen Diller Family Comprehensive Cancer Center
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000463168; UCSF-02257; UCSF-2214; UCSF-H24045-22163-04
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-10

CONDITIONS: Anemia; Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; adult acute lymphoblastic leukemia in remission; recurrent adult lymphoblastic lymphoma; anemia; refractory chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; Waldenstrom macroglobulinemia; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma; polycythemia vera; essential thrombocythemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; relapsing chronic myelogenous leukemia; chronic eosinophilic leukemia; chronic idiopathic myelofibrosis; chronic myelomonocytic leukemia; chronic neutrophilic leukemia; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult acute lymphoblastic leukemia; stage I multiple myeloma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Anemia; Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Congenital Abnormalities; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Polycythemia Vera; Thrombocythemia, Essential; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic | interventions — Filgrastim; Busulfan; fludarabine phosphate; Methotrexate; Tacrolimus; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: busulfan
Drug: fludarabine phosphate
Drug: methotrexate
Drug: tacrolimus
Procedure: allogeneic bone marrow transplantation
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as busulfan and fludarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy with a peripheral stem cell or bone marrow transplant may allow more chemotherapy to be given so that more cancer cells are killed. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Tacrolimus and methotrexate may stop this from happening.

PURPOSE: This phase II trial is studying how well giving busulfan together with fludarabine before donor stem cell transplant works in treating patients with hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety, in terms of treatment-related mortality at 100 days post-transplantation, of a myeloablative preparative regimen comprising busulfan and fludarabine and graft-vs-host disease (GVHD) prophylaxis comprising tacrolimus and methotrexate in patients with hematopoietic disorders undergoing matched unrelated donor stem cell transplantation.
* Determine the efficacy, in terms of overall survival at 1-year post-transplantation, in patients treated with this regimen.

Secondary

* Determine organ toxicity in patients treated with this regimen.
* Determine neutrophil and platelet recovery in patients treated with this regimen.
* Determine the incidence and severity of acute and chronic GVHD in patients treated with this regimen.

OUTLINE:

* Myeloablative preparative regimen: Patients receive busulfan IV over 2 hours every 6 hours on days -7 to -4 and fludarabine IV over 30 minutes on days -7 to -3.
* Allogeneic stem cell transplantation: Patients undergo allogeneic peripheral blood stem cell or bone marrow transplantation on day 0. Patients also receive filgrastim (G-CSF) subcutaneously daily beginning on day 7 and continuing until blood counts recover.
* Graft-vs-host disease prophylaxis: Patients receive tacrolimus IV continuously beginning on day -2 and continuing until discharged from the hospital (may convert to oral dosing administered twice daily when tolerated) and methotrexate IV over 15-30 minutes on days 1, 3, 6, and 11.

After completion of study therapy, patients are followed periodically.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following hematopoietic disorders:

  * Chronic myelogenous leukemia (CML), meeting 1 of the following criteria:

    * Chronic phase disease failing imatinib mesylate therapy

      * Progressive disease OR failed to achieve a major cytogenetic response at 1 year after initiation of therapy
    * Accelerated phase disease, meeting 1 of the following criteria:

      * Failed to achieve complete cytogenetic remission at 1 year after initiation of therapy
      * Failed to achieve any cytogenetic response at 3 or 6 months during therapy
      * Progressive disease, demonstrated by worsening cytogenetic response in 2 consecutive analyses separated by 4 weeks
    * Blast crisis with < 10% blasts in bone marrow within 6 weeks of transplantation
  * Acute myeloid leukemia (AML), meeting 1 of the following criteria:

    * In second or greater remission
    * In first remission with poor prognosis cytogenetics [-5, -5q, -7, -7q and ≥ 2 cytogenetic abnormalities, t(6,9), t(9,11), or Philadelphia chromosome]
    * In hematologic remission but with persistent cytogenetic abnormalities
    * Primary refractory AML with < 10% blasts in bone marrow within 6 weeks of transplantation
  * Myelodysplasia with < 20% blasts in bone marrow within 6 weeks of transplantation and meeting 1 of the following criteria:

    * Advanced disease (International Prognostic Scoring System [IPSS] score intermediate-1, intermediate-2, or high risk)
    * Myelodysplastic syndromes (MDS) with progression to AML
    * Treatment-related AML
  * Acute lymphocytic leukemia (ALL), meeting 1 of the following criteria:

    * In second or greater remission
    * In first remission with high-risk cytogenetics [Philadelphia chromosome; t(4,11); and -7]
    * Primary refractory ALL with < 10% blasts in the bone marrow
  * Severe aplastic anemia that has failed immunosuppressive therapy
  * Non-Hodgkin's lymphoma, meeting 1 of the following criteria:

    * In second or greater remission
    * Relapsed disease in a patient not eligible for autologous stem cell transplantation
  * Lymphoproliferative disease (e.g., chronic lymphocytic leukemia or Waldenstrom's macroglobulinemia), meeting 1 of the following criteria:

    * In second or greater remission
    * Relapsed disease in a patient not eligible for autologous stem cell transplantation
  * Multiple myeloma, meeting 1 of the following criteria:

    * Stage II or III disease in first or greater relapse
    * Refractory disease
    * Newly diagnosed disease with chromosome 13 abnormalities
  * Advanced myeloproliferative disease, meeting 1 of the following criteria:

    * Myelofibrosis requiring > 2 units of packed red blood cells each month
    * Essential thrombocythemia or polycythemia rubra vera that has progressed to AML
    * Failed prior AML therapy
* No active, uncontrolled CNS leukemia
* Not eligible for autologous or mini-allogeneic transplantation
* No fully matched or single-antigen mismatched sibling donor available
* HLA-matched unrelated donor available

  * HLA typed at HLA-A, -B, -C, -DRB1 and/or -DQB1 by high-resolution techniques
  * For patients without HLA identical donors, mismatches at DQ (i.e., 8/8 match) and 1 additional mismatch at the allele level at HLA-A, -B, -C, or -DRB1 (i.e., 7/8 molecular match) allowed

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Creatinine < 2.0 mg/dL
* Pulmonary diffusing capacity > 40% of predicted
* Cardiac ejection fraction > 40% by MUGA or echocardiography
* No active liver disease
* Bilirubin ≤ 2.0 mg/dL
* Alkaline phosphatase < 3 times upper limit of normal (ULN)
* AST < 3 times ULN
* Hepatitis C or active hepatitis B (HBV) allowed provided a liver biopsy is performed and ≤ grade 2 inflammation is present

  * Patients with active HBV viral replication must receive antiviral therapy
* HIV negative
* No ongoing active infection
* Not pregnant or nursing
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 3 weeks since prior chemotherapy except for hydroxyurea or imatinib mesylate
* More than 3 months since prior interferon

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2002-01; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Treatment-related mortality in the first 100 days post-transplant
Overall survival at 1 year post-transplant

SECONDARY OUTCOMES:
Incidence and severity of organ-specific toxicity
Engraftment including neutrophil and platelet recovery and donor chimerism at 3 and 12 months post-transplant
Rate of acute graft-vs-host disease (GVHD)
Rate of chronic GVHD

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G. Martin, MD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States